CLINICAL TRIAL: NCT06726382
Title: KF2024#1-trial: Esketamine Interaction Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Janne Backman, Professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KF2024#1; 2024-516892-34-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-03; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Drug Interactions; Food-drug Interaction
MeSH Terms: interventions — Esketamine; Cobicistat; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Esketamine Nasal Spray (Active Comparator): 250 ml water at 8.00 and 9.00 a.m. on the study day. Study drug dose (Esketamine Spravato, 28 mg) nasally at 9.00 a.m. on the study day.
  Interventions: Drug: Esketamine Nasal Spray
- Esketamine p.o. and water (Experimental): 250 ml water at 8.00 and 9.00 a.m. on the study day. Study drug dose (Esketamine Kalceks 5 mg/ml, 28 mg) p.o. at 9.00 a.m. on the study day.
  Interventions: Drug: Esketamine 28 mg
- Esketamine p.o. and grapefruit juice (Experimental): 250 ml grapefruit juice at 8.00 and 9.00 a.m. on the study day. Study drug dose (Esketamine Kalceks 5 mg/ml, 28 mg) p.o. at 9.00 a.m. on the study day.
  Interventions: Drug: Esketamine 28 mg
- Esketamine p.o. and Cobisistat (Experimental): 150 mg Cobisistat and 250 ml water at 8.00 a.m. on the study day. Study drug dose (Esketamine Kalceks 5 mg/ml, 28 mg) p.o. and 250 ml water at 9.00 a.m. on the study day.
  Interventions: Drug: Esketamine 28 mg; Drug: Cobicistat 150 MG

INTERVENTIONS:
Drug: Esketamine Nasal Spray — 1 x 28 mg dose
  Other Names: Esketamine, Spravato, Janssen-Cilag International NV
  Arms: Esketamine Nasal Spray
Drug: Esketamine 28 mg — 1 x 5,6 ml p.o.
  Other Names: Esketamine Kalceks 5 mg/ml, AS KALCEKS
  Arms: Esketamine p.o. and Cobisistat; Esketamine p.o. and grapefruit juice; Esketamine p.o. and water
Drug: Cobicistat 150 MG — 1 x 150 mg tablet
  Other Names: Tybost 150 mg tablet, GILEAD
  Arms: Esketamine p.o. and Cobisistat

SUMMARY:
Esketamine is a drug which is used for depression treatment, to relieve pain and, in larger doses, in anesthesia. Spravato nasal spray is the only esketamine product on the market used for the treatment of depression, but the high price limits the use of the drug.

The aim of this study is to compare the concentration of esketamine after nasal (licensed product Spravato) and oral administration with and without a CYP3A4 inhibitor. Grapefruit juice and cobicistat are studied as CYP3A4 inhibitors in the study.

In an open four-phase, randomized, alternating study with 12 healthy volunteers, the subjects will receive Spravato 28 mg nasal or esketamine 28 mg oral with either grapefruit juice, cobicistat or water in the study facilities. Blood samples will be collected and esketamine pharmacokinetics will be monitored up to 24 hours postdose. Primary endpoint is area under the plasma concentration-time curve of esketamine.

ELIGIBILITY:
Inclusion Criteria:

* signed consent
* age 18-45 years
* healthy
* no indications of substance abuse
* Accepted results from laboratory tests (blood hemoglobin, basic blood count and blood platelets, alanine aminotransferase, alkaline phosphatase, glutamyl transferase, creatinine, plasma potassium and sodium). Negative pregnancy test result (serum human chorionic gonadotropin) for women.
* no significant abnormalities in the ECG
* systolic blood pressure 140 mmHg-100 mmHg
* heart rate ≥50/minute

Exclusion Criteria:

* significant illness
* less than 3 months since the last clinical trial
* less than 3 months after donating blood
* significant overweight/poor veins
* BMI below 18.5 kg/m2
* past or present mood disorder or suicidality
* substance abuse
* systolic blood pressure below 100 mmHg or above 140 mmHg
* heart rate <50/minute
* conduction disorder or other significant abnormality in the ECG
* smoking
* regular medication (including e-pills and other preparations containing estrogens)
* pregnancy or its planning or breastfeeding
* hypersensitivity to investigational drugs or excipients of medicinal products
* use of natural products (such as St. John's wort)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration - time curve of esketamine | Prior to and 10, 20, 30, 40, 50, 60, 75, 90, 105 min and 2 , 3, 4, 6, 8, 10, 12 and 24 hours after administration the drug.

SECONDARY OUTCOMES:
Peak plasma concentration for both esketamine and its metabolites | Prior to and 10, 20, 30, 40, 50, 60, 75, 90, 105 min and 2 , 3, 4, 6, 8, 10, 12 and 24 hours after administration the drug.
Half-life for both esketamine and its metabolites | Prior to and 10, 20, 30, 40, 50, 60, 75, 90, 105 min and 2 , 3, 4, 6, 8, 10, 12 and 24 hours after administration the drug.
Time to peak plasma concentration for both esketamine and its metabolites | Prior to and 10, 20, 30, 40, 50, 60, 75, 90, 105 min and 2 , 3, 4, 6, 8, 10, 12 and 24 hours after administration the drug.
Fractional areas under concentration-time curve (AUC) for both esketamine and its metabolites | Prior to and 10, 20, 30, 40, 50, 60, 75, 90, 105 min and 2 , 3, 4, 6, 8, 10, 12 and 24 hours after administration the drug.
Areas under concentration-time curve (AUC) for esketamine metabolites | Prior to and 10, 20, 30, 40, 50, 60, 75, 90, 105 min and 2 , 3, 4, 6, 8, 10, 12 and 24 hours after administration the drug.
Blood pressure | 0, 60, 120 and 240 min after administration
  Blood pressure (safety parameter)
Heart rate | 0, 60, 120 and 240 min after administration
  Heart rate (Safety parameter)

CONTACTS AND LOCATIONS:
Overall Officials: Janne T Backman, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Department of Clinical Pharmacology, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No